CLINICAL TRIAL: NCT03897361
Title: A Phase 1/2 Study to Determine Safety and Efficacy of Transplantation With Autologous Human CD34+ Hematopoietic Stem Cells (HSC) From Mobilized Peripheral Blood Stem Cells (PBSC) of Patients With Cystinosis Modified by Ex Vivo Transduction Using pCCL-CTNS or pCDY.EFS.CTNS.T260I Lentiviral Vector and Will Include Transduction Enhancer When Required During Manufacturing
Brief Title: Stem Cell Gene Therapy for Cystinosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other); Cystinosis Research Foundation (Other)
Responsible Party: Principal Investigator, Stephanie Cherqui, Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 018631
Record Dates: First submitted 2019-02-06; First posted 2019-04-01 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-08

CONDITIONS: Lysosomal Storage Diseases; Cystinosis
Keywords: Cystinosis; Lysosomal Storage Disorders; LSD
MeSH Terms: conditions — Lysosomal Storage Diseases; Cystinosis

STUDY DESIGN:
Intervention Model Description: This study will include up to 6 subjects and follows a 3-cohort staggered treatment design with 2 subjects per cohort. The first 2 cohorts will consist of 4 adults (18 years or older), potentially followed by a cohort consisting of 2 adolescents or adults (>14 years old).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gene Therapy with CTNS-RD-04 or CTNS-RD-04-LB (where the suffix "-LB" stands for LentiBOOST) (Experimental): This is a single arm study without randomization. Eligible subjects will receive the final product: CTNS-RD-04 or CTNS-RD-04-LB (where the suffix "-LB" stands for LentiBOOST).
  Interventions: Genetic: CTNS-RD-04 or CTNS-RD-04-LB (where the suffix "-LB" stands for LentiBOOST)

INTERVENTIONS:
Genetic: CTNS-RD-04 or CTNS-RD-04-LB (where the suffix "-LB" stands for LentiBOOST) — Peripheral blood autologous CD34+ enriched cell fraction transduced with lentiviral vector, pCCL-CTNS or pCDY.EFS.CTNS.T260I, that contains the human CTNS complementary deoxyribonucleic acid (cDNA) sequence.

SUMMARY:
This study is a Phase 1/2 clinical trial that will assess the safety and efficacy of enriched gene-corrected hematopoietic stem cells isolated from patients affected with cystinosis. (Investigational Product: CTNS-RD-04 or CTNS-RD-04-LB, where the suffix "-LB" stands for LentiBOOST)

DETAILED DESCRIPTION:
Cystinosis is a rare inherited recessive disease belonging to the family of Lysosomal Storage Disorders and is characterized by lysosomal accumulation of cystine in all the cells of the body leading to multi-organ failure. Cystinosis has a devastating impact on the affected individuals, primarily children, and young adults, even with cysteamine treatment. The prevalence of cystinosis is 1 in 100,000 to 1 in 200,000. The gene involved in cystinosis is the gene CTNS that encodes for the transmembrane lysosomal cystine transporter - cystinosin. The current standard of care does not prevent the progression of the disease and significantly impacts the quality of life of patients with cystinosis.

For this study, up to 6 subjects meeting eligibility criteria will be transplanted following a 3-cohort staggered treatment design with 2 subjects per cohort. The first 2 cohorts will consist of 4 adults (18 years or older), potentially followed by a cohort consisting of 2 adolescents or adults (> 14 years old). Following the informed consent process, enrolled subjects will be screened to confirm full eligibility for participation. Eligible subjects will undergo hematopoietic stem cell (HSC) mobilization and collection (leukapheresis). A portion of cells will be kept as "back-up" for rescue purpose if necessary, and a portion will be ex vivo gene-modified with a lentiviral vector, pCCL-CTNS or pCDY.EFS.CTNS.T260I, to express CTNS gene (product name: CTNS-RD-04). Clinical manufacturing for patients in Cohort 3 will introduce a transduction enhancer LentiBOOST (product name for these patients will be CTNS-RD-04-LB, where the suffix "-LB" stands for LentiBOOST). The subjects will receive marrow cytoreduction with busulfan prior to infusion of CTNS-RD-04. Subjects will discontinue cysteamine treatment during the assessment period. The assessment follow-up period will include an initial 2 years of active end-point evaluations, where the subjects will be evaluated at 3-, 6-, 9-, 12-, 18- and 24-months post-transplantation. A Long-Term Follow-Up study (LTFU) for a total 15-year follow-up period will be offered to all subjects.

The objectives of this Phase 1/2 clinical study are to assess the safety/tolerability of CTNS-RD-04, and its efficacy through a number of clinical, molecular and biochemical assessments.

ELIGIBILITY:
Inclusion Criteria:

The following criteria must be met by all subjects considered for study participation.

1. Cohorts 1 and 2: Male or female subject is ≥ 18 years of age.
2. Cohort 3: Male or female subject is ≥ 14 years of age.
3. Subject is diagnosed with cystinosis, i.e., early onset of Fanconi syndrome, and history of elevated white blood cell cystine level and/or history of or presence of cystine crystals in the eye.
4. Subject has a Karnofsky Performance Status or age-dependent Lansky Performance of ≥ 60.
5. If subject has had a kidney transplant, he or she must be at least one-year post kidney transplant status.
6. Subject has adequate hematologic function:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 1000/mm^3
   2. Platelet count ≥ 100 x 1000/mm^3
   3. Hemoglobin ≥ 9.0 gm/dL
7. Subject has an adequate hepatic function:

   1. Bilirubin ≤ 2.0 mg/ dL
   2. ALT ≤ 3 x institution's upper limit of normal (ULN) U/L
8. Subject has an adequate renal function:

   a. Serum creatinine <2x ULN mg/dL
9. Subject has adequate coagulation:

   1. PT/aPTT ≤ 1.2 x ULN seconds
   2. INR ≤ 2
10. Subject has adequate thyroid function (with or without thyroid replacement therapy):

    1. TSH 0.27-4.2 mIU/mL
    2. Total T4 ≤ 2 x ULN mcg/dL
11. If female: female of childbearing potential (i.e., not surgically sterile [tubal ligation, hysterectomy, or bilateral oophorectomy] or not at least 2 years naturally postmenopausal) agrees to remain sexually abstinent or utilize the same acceptable form of highly effective contraception from screening through two years post-transplant.

    The acceptable forms of contraception for this study include hormonal contraceptives (oral, implant, transdermal patch, or injection) associated with inhibition of ovulation at a stable dose for at least 3 months prior to screening, barrier (condom with spermicide, diaphragm with spermicide), intrauterine device, or a partner who has been vasectomized for at least 6 months and has documented medical assessment of surgical success of a vasectomy.

    Note: males with cystinosis are sterile.
12. If male: males must agree to remain sexually abstinent or utilize an acceptable form of highly effective contraception from screening through two years post-transplant.
13. Subject is willing and able to comply with the study restrictions and requirements.
14. Subject is willing to provide written informed consent/permission/assent prior to participation in the study.
15. Subject must be willing to refrain from donating sperm after receiving the conditioning regimen. For subjects planning on (or for whom there is a possibility of) fathering children in the future, sperm banking prior to administration of conditioning regimen will be recommended.
16. Subject must be willing to refrain from donating blood, organs, tissues, or cells for transplantation from 30 days prior to screening through any time after CTNS-RD-04 treatment.
17. Subject must be willing and must be able (in the judgment of the investigator) to discontinue his or her cysteamine therapy (oral and/or eye drop).

Exclusion Criteria:

1. Subject has an active, uncontrolled, acute bacterial, viral, or fungal infection during screening or within 30 days prior to starting the conditioning regimen.
2. Subject has positive serology at screening for any of the following:

   1. Human Immunodeficiency Virus (HIV) 1-2
   2. Human T-cell Lymphotropic Virus (HTLV) - I/II
   3. Hepatitis B core and Hepatitis B PCR positive
   4. Hepatitis C Virus (HCV)
   5. Rapid Plasma Reagin (RPR)
   6. Chagas' Disease (T. curzi)
   7. QuantiferonTB
   8. Nucleic Acid Test (NAT) for HIV
   9. West Nile Virus (WNV)
3. Subject has a known clinically significant immunodeficiency disorder.
4. Subject is a female of childbearing potential that is nursing, planning a pregnancy or has a positive serum pregnancy test.
5. Subject has received a prior marrow or stem cell transplantation or is planning to receive one within 90 days of study initiation.
6. Subject has had an active bleeding disorder within 90 days prior to screening OR requires anticoagulation therapy prior to treatment with ex vivo gene therapy.
7. Subject has an active malignancy or history of malignancy including lymphoma (except primary, cutaneous basal cell or squamous cell cancer appropriately treated prior to transplantation).
8. Subject has an end-stage renal disease (defined as GFR <15 mL/min) and is already on a transplantation list or who may be planning to register for a kidney transplant within 90 days of study initiation.
9. Subject has impaired pulmonary function (based on FEV1 of <=50% of predicted or DLCO of <=40 % of predicted and gender-specific normal threshold value).
10. Subject has impaired cardiac function within 90 days prior to screening including any of the following:

    1. Myocardial infarction
    2. Clinically significant abnormal electrocardiogram (ECG)
    3. Ejection fraction of < 40%
    4. Uncontrolled arrhythmia
    5. Other clinically significant heart disease (e.g., congestive heart failure, uncontrolled hypertension, history of labile hypertension).
11. Subject has a severe or uncontrolled medical disorder (e.g., pancreatitis, severe liver disease, unstable diabetes mellitus) that would, in the investigators' opinion, impair their ability to receive study treatment and follow the study procedures.
12. Subject has a history of allergic reactions attributed to compounds of similar chemical or biologic composition to Busulfan or allergy or contraindication to use of other agents used in the study, including iohexol, acid-citrate-dextrose Formula A (ACDA), G-CSF or plerixafor.
13. Subject has a known history of drug or alcohol addiction.
14. Subject has undergone major surgery within 90 days (or longer if not fully recovered) prior to screening.
15. Subject is receiving cytotoxic or immunosuppressive agents, other than for kidney transplant, within 60 days prior to screening or requires treatment with such agents prior to treatment with ex vivo gene therapy.
16. Subject has previously received gene therapy at any time.
17. Subject is currently receiving or anticipates receiving another investigational agent, device, or procedure from 30 days prior to screening through study completion.
18. Subject has any condition, in the opinion of the investigator, that compromises compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-18 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: Total number of adverse events (AEs) per participant (pre- and post-dose to end of study) | From the first pre-dose safety visit to the end of the treatment period (e.g., 24 months post-dose) or the participant's last safety-assessment visit, whichever occurs later.
  The total count of all adverse events (AEs) recorded for each dosed participant reported at any scheduled study visit starting with the first pre-dose safety visit (i.e., the first visit after informed consent and before the first administration of study drug) and continuing through the end of the treatment period. Events were coded using MedDRA v24.0. The outcome is the total count of AEs per participant. Excludes ongoing AEs at end of study that are captured in separate long-term follow-up study.
  Unit of Measure: Count (events per participant)
Safety and tolerability: Aggregate number of adverse events (AEs) by National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) severity (pre-dose and post-dose to end of study) | From the first pre-dose safety visit to the end of the treatment period (e.g., 24 months post-dose) or the participant's last safety-assessment visit, whichever occurs later.
  The total aggregate count of all graded adverse events (AEs) recorded for all dosed participants reported at any scheduled study visit starting with the first pre-dose safety visit (i.e., the first visit after informed consent and before the first administration of study drug) and continuing through the end of the treatment period. Events were coded using MedDRA v24.0 and graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. The outcome is the total count of AEs per grade (Mild, Moderate, Severe, Life Threatening, Death). Excludes ongoing AEs at end of study that are captured in separate long-term follow-up study.
  Unit of Measure: Count (events) - separate counts for each CTCAE grade.
Safety and tolerability: Aggregate number of adverse events (AEs) by relationship to study treatment (pre-dose and post-dose to end of study) | From the first pre-dose safety visit to the end of the treatment period (e.g., 24 months post-dose) or the participant's last safety-assessment visit, whichever occurs later.
  The total aggregate count of all adverse events (AEs) categorized by relationship to the study treatment recorded for all dosed participants reported at any scheduled study visit starting with the first pre-dose safety visit (i.e., the first visit after informed consent and before the first administration of study drug) and continuing through the end of the treatment period. Relationship to the study treatment was determined using the standard categories defined in the protocol: • Related (probably or possibly related) • Unrelated (not related, unlikely related). Each AE was coded with MedDRA v24.0. The outcome reported is the study-wide total count of AEs in each relationship category. Excludes ongoing AEs at end of study that are captured in separate long-term follow-up study.
  Unit of Measure: Count (events) - separate counts for each relationship category (Related, Unrelated)
Safety and tolerability: Clinical laboratory values for white blood cell, absolute monocyte, and platelet counts at baseline, 12 month and 24 month post-infusion study visits reported at individual participant level. | Baseline, 12 months post-infusion, 24 months post-infusion
  Clinical laboratory values for white blood cell, absolute monocyte, and platelet counts at baseline, 12 month and 24 month post-infusion study visits. No summary statistics will be reported - each participant-level value will be uploaded as individual participant data.
  Unit of Measure: White blood cell count (1000/mmHg^3), Absolute monocyte count (1000/mmHg^3), Platelet count (1000/mmHg^3) where mmHG^3 is millimeters of mercury cubed- raw individual values
Safety and tolerability: Systolic and diastolic blood pressure at baseline, 12 month and 24 month post-infusion study visits reported at individual participant level. | Baseline, 12 months post-infusion, 24 months post-infusion
  Systolic and diastolic blood pressure at baseline, 12 month and 24 month post-infusion study visits. Measurement taken with the subjects positioned supine, seated or semi-fowlers. No summary statistics will be reported - each participant-level value will be uploaded as individual participant data.
  Unit of Measure: blood pressure in millimeters of mercury (mmHg) - raw individual values
Safety and tolerability: Heart rate at baseline, 12 month and 24 month post-infusion study visits reported at individual participant level. | Baseline, 12 months post-infusion, 24 months post-infusion
  Heart rate at baseline, 12 month and 24 month post-infusion study visits. Measurement taken with the subjects positioned supine, seated or semi-fowlers. No summary statistics will be reported - each participant-level value will be uploaded as individual participant data.
  Unit of Measure: beats per minute (BPM) - raw individual values
Safety and tolerability: Body temperature at baseline, 12 month and 24 month post-infusion study visits reported at individual participant level. | Baseline, 12 months post-infusion, 24 months post-infusion
  Body temperature at baseline, 12 month and 24 month post-infusion study visits. No summary statistics will be reported - each participant-level value will be uploaded as individual participant data.
  Unit of Measure: degrees Celsius - raw individual values
Safety and tolerability: Respiratory rate at baseline, 12 month and 24 month post-infusion study visits reported at individual participant level. | Baseline, 12 months post-infusion, 24 months post-infusion
  Respiratory rate at baseline, 12 month and 24 month post-infusion study visits. Measurement taken with the subjects positioned supine, seated or semi-fowlers. No summary statistics will be reported - each participant-level value will be uploaded as individual participant data.
  Unit of Measure: breaths per minute - raw individual values
Safety and tolerability: Electrocardiogram (ECG) ventricular rates at baseline, 12 month and 24 month post-infusion study visits reported at individual participant level. | Baseline, 12 months post-infusion, 24 months post-infusion
  Electrocardiogram (ECG) ventricular rates at baseline, 12 month and 24 month post-infusion study visits. ECG recordings will be obtained using standard 12-lead resting ECGs with a bandwidth of 0.05-100 Hz and a minimum sampling rate of 500 Hz. No summary statistics will be reported - each participant-level value will be uploaded as individual participant data.
  Unit of Measure: ECG beats per minute (BPM) - raw individual values
Safety and tolerability: Electrocardiogram (ECG) intervals including PR interval, QRS interval, QT interval and QTc Bazett at baseline, 12 month and 24 month post-infusion study visits reported at individual participant level. | Baseline, 12 months post-infusion, 24 months post-infusion
  Electrocardiogram (ECG) intervals including PR interval, QRS interval, QT interval and QTc Bazett at baseline, 12 month and 24 month post-infusion study visits. ECG recordings are obtained using standard 12-lead resting ECGs with a bandwidth of 0.05-100 Hz and a minimum sampling rate of 500 Hz. No summary statistics will be reported - each participant-level value will be uploaded as individual participant data.
  Unit of Measure: ECG Intervals in milliseconds (ms) - raw individual values
Safety: Number of dosed participants showing evidence (positive or negative) of genotoxicity as determined by polyclonal expansion and insertional mutagenesis. | Up to 24 months post transplant.
  Number of dosed participants that show evidence (positive or negative) of polyclonal expansion and insertional mutagenesis as measured in whole blood collected at several timepoints throughout the study (Baseline, 1-, 3-, 6-, 12-, 18-, 24-, months post-transplant) using vector integration site (VIS) analysis. VIS is performed through LTR-based PCR amplification and Illumina sequencing. Clonal abundance is monitored using the Sonic Abundance method.
  Unit of Measure: Participants

SECONDARY OUTCOMES:
Efficacy: Cystine levels in leukocytes and granulocytes at baseline, 12 month and 24 month post-infusion study visits reported at individual participant level. | Baseline, 12 months post-infusion, 24 months post-infusion.
  Cystine levels in leukocytes and granulocytes from whole blood collected at baseline, 12 month and 24 month post-infusion study visits. Liquid chromatography tandem mass spectrometry (LC-MS/MS), using d4-cystine as an internal standard is used to measure cystine levels. No summary statistics will be reported - each participant-level value will be uploaded as individual participant data.
  Unit of measure: nanomole half-cystine per milligram protein (nmol half-cystine per mg protein) - raw individual values
Efficacy: Clinical laboratory values of estimated glomerular filtration rate (eGFR) at baseline, 12 month and 24 month post-infusion study visits reported at individual participant level. | Baseline, 12 months post-infusion, 24 months post-infusion
  Renal glomerular and tubular function: Clinical laboratory values of creatinine in whole blood collected at baseline, 12 month and 24 month post-infusion study visits are used to calculate corresponding estimated glomerular filtration rate (eGFR) using the 2021 CKD-EPI equation. No summary statistics will be reported - each participant-level value will be uploaded as individual participant data.
  Unit of measure: milliliters per minute per 1.73 meters squared (mL/min/1.73m^2) - raw individual values
Efficacy: Clinical laboratory values of thyroxine (T4) endocrine levels at baseline, 12 month and 24 month post-infusion study visits reported at individual participant level. | Baseline, 12 months post-infusion, 24 months post-infusion
  Endocrine function: Clinical laboratory values of thyroxine (T4) hormone levels from whole blood collected at baseline, 12 month and 24 month post-infusion study visits. No summary statistics will be reported - each participant-level value will be uploaded as individual participant data.
  Unit of measure: Unit of measure: units per deciliter (ud/dL) - raw individual values
Efficacy: Clinical laboratory values thyroid-stimulating hormone (TSH) endocrine levels at baseline, 12 month and 24 month post-infusion study visits reported at individual participant level. | Baseline, 12 months post-infusion, 24 months post-infusion
  Endocrine function: Clinical laboratory values of thyroid stimulating hormone (TSH) levels from whole blood collected at baseline, 12 month and 24 month post-infusion study visits. No summary statistics will be reported - each participant-level value will be uploaded as individual participant data.
  Unit of measure: micro-international units per milliliter (uIU/mL) - raw individual values
Transduction Efficiency: Vector copy number (VCN) in peripheral blood at 12 month and 24 month post-infusion study visits reported at individual participant level. | 12 months post-infusion and 24 months post-infusion
  Evaluation of engraftment and gene transcription (transduction efficiency) will be assessed by measuring vector copy number (VCN) in peripheral blood cells extracted from participant whole blood collected at 12 month and 24 month post-transplant. ddPCR of particpant peripheral blood cells and a transduced and non-transduced control are used in each VCN assay. No summary statistics will be reported - each participant-level value will be uploaded as individual participant data.
  Unit of measure: Vector Copy Number per diploid genome (VCN/dg) - raw individual values

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Cherqui, Ph.D., Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending [5] years following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.

REFERENCES:
- [Result] Harrison F, Yeagy BA, Rocca CJ, Kohn DB, Salomon DR, Cherqui S. Hematopoietic stem cell gene therapy for the multisystemic lysosomal storage disorder cystinosis. Mol Ther. 2013 Feb;21(2):433-44. doi: 10.1038/mt.2012.214. Epub 2012 Oct 23. PMID 23089735
- [Result] Naphade S, Sharma J, Gaide Chevronnay HP, Shook MA, Yeagy BA, Rocca CJ, Ur SN, Lau AJ, Courtoy PJ, Cherqui S. Brief reports: Lysosomal cross-correction by hematopoietic stem cell-derived macrophages via tunneling nanotubes. Stem Cells. 2015 Jan;33(1):301-9. doi: 10.1002/stem.1835. PMID 25186209